CLINICAL TRIAL: NCT03851861
Title: Dietary Intervention and Gastrointestinal Function in Patients With Parkinson's Disease
Acronym: MED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201900252; OCR20178 (Other: UF OnCore)
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease
Keywords: Intestinal Permeability; Mediterranean Diet; Leaky Gut; Intestinal Barrier Function
MeSH Terms: conditions — Parkinson Disease | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: A prospective intervention study in which participants with diagnosed Parkinson's disease are instructed to follow the Mediterranean diet for a 5-week intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mediterranean Diet (Experimental): Participants will be given individualized diet education on the Mediterranean diet and instructed to follow the diet for the 5-week intervention period. Individualized diet education will be administered by a licensed, registered dietitian nutritionist (RDN) followed by weekly phone calls to ensure compliance, improve adherence to the diet and monitor for adverse events.
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Mediterranean Diet — Participants will be instructed to include the following in their diet: a) abundant use of olive oil for cooking and dressing dishes; b) consumption of ≥2 daily servings of vegetables; c) ≥2-3 daily serving of fresh fruits (including natural juices); d) ≥3 weekly servings of legumes; e) ≥3 weekly servings of fish or seafood (at least one serving of fatty fish); f) ≥3 weekly serving of nuts or seeds; g) select white instead of red meats or processed meats (burgers, sausages); h) cook at least twice a week with a tomato herb sauce.
  Participants will be instructed to eliminate or limit the consumption of the following foods: cream, butter, margarine, cold meat, paté, duck, carbonated and/or sugared beverages, pastries, industrial bakery products and desserts, French fries or potato chips, and out-of-home pre-cooked cakes and sweets. For usual drinkers, the main source of alcohol should be wine.

SUMMARY:
In this prospective, intervention study, participants with diagnosed Parkinson's disease will be instructed to follow a Mediterranean diet for five weeks. Gut permeability will be assessed using food-grade sugar molecules. Participants will provide urine and stool samples to assess gut permeability and microbial communities.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed Parkinson's disease aged 21-85 years
* Hoehn & Yahr stage <3
* Currently living in the same household with a healthy spouse/partner who meets study eligibility criteria and is willing to participate
* Willing and able to complete informed consent in English
* Willing to complete daily and weekly questionnaires and 6 dietary recalls over approximately 7 weeks
* Willing to avoid beer, wine, and cocktails on the day before and the day of the sugar probe tests.
* Willing to provide urine and stool samples during the study collection periods.
* Willing and able to fast (no food or drink, except water or tea) for a prolonged period of time during study urine collections.
* Willing to maintain usual diet through the pre-baseline period
* Willing to make dietary changes to follow a Mediterranean dietary pattern during the intervention period.
* Willing to discontinue taking prebiotic, fiber, probiotic, herbal, or high-dose vitamin or mineral supplements that may impact inflammation during the pre-baseline period and throughout the study protocol.
* Willing to limit use of oral laxative medication to an "as-needed basis" (i.e. <3 times per week) during the full length of the study
* Willing to avoid high intensity exercises two days prior to and the day of the permeability tests. These tests will be done on two occasions.
* Willing to provide a social security number to receive study payment.

Exclusion Criteria:

* Does not meet above criteria
* Atypical or secondary Parkinsonism
* History of deep brain stimulation
* Daily use of NSAIDs in the last 3 months or incidental use in the last 2 weeks prior to screening.
* Daily use of anticholinergics or prokinetic agents
* Use of enemas or suppositories to alleviate constipation
* Use of another investigational product within 3 months of the screening visit.
* Antibiotic use within 2 months from the day of stool collection
* Good adherence to the Mediterranean diet during the pre-baseline period (score >6) based on the 14-item Mediterranean Diet Assessment Tool
* Physician-diagnosed gastrointestinal disease or condition (such as ulcerative colitis, Crohn's disease, gastroparesis, cancer, peptic ulcer disease, Celiac disease, short bowel disease, ileostomy, colostomy) other than gastroesophageal reflux or diverticular disease

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Gastroduodenal Permeability | Week 1; Week 5
  The primary outcome is the change in gastroduodenal permeability induced by the Mediterranean diet. Gastroduodenal permeability will be assessed by measuring sucrose concentration in the 0 to 5-hour urine collection (end of intervention minus baseline)

SECONDARY OUTCOMES:
Small Intestinal Permeability | Week 1; Week 5
  The change in lactulose/rhamnose concentrations in a 5-hour urine collection (end of intervention minus baseline)
Colonic Permeability | Week 1; Week 5
  The change in sucralose/erythritol concentrations in a 5 to 24 hour urine collection (end of intervention minus baseline)
Whole Gut Permeability | Week 1; Week 5
  The change in sucralose/erythritol concentrations in a 0 to 24 hour urine collection (end of intervention minus baseline)
Stool Frequency | Week 1; Week 5
  Difference in the average number of weekly stools (end of intervention compared to baseline)
Stool Consistency | Week 1; Week 5
  Daily GI symptoms assessed using the Bristol Stool Scale (BSS). Difference in the average BSS (end of intervention compared to baseline).
Gastrointestinal Symptoms | Week 1; Week 5
  Weekly GI symptoms assessed using the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS consists of 15 questions related to 5 syndromes, constipation, diarrhea, reflux, abdominal pain, and indigestion. Symptoms are scored 1=no discomfort to 7=very severe discomfort. Scores from each of the 15 questions are summed for the total GSRS score.

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — Univeristy of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rusch C, Beke M, Tucciarone L, Nieves C Jr, Ukhanova M, Tagliamonte MS, Mai V, Suh JH, Wang Y, Chiu S, Patel B, Ramirez-Zamora A, Langkamp-Henken B. Mediterranean Diet Adherence in People With Parkinson's Disease Reduces Constipation Symptoms and Changes Fecal Microbiota After a 5-Week Single-Arm Pilot Study. Front Neurol. 2021 Dec 23;12:794640. doi: 10.3389/fneur.2021.794640. eCollection 2021. PMID 35002935